CLINICAL TRIAL: NCT03019198
Title: TRANEXAMIC ACID IN PATIENTS UNDERGOING TOTAL HIP ARTHROPLASTY IN A BRAZILIAN REFERENCE ORTHOPEDIC CENTER: A RANDOMIZED CONTROLLED TRIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Traumatologia e Ortopedia (Other Government)
Responsible Party: Principal Investigator, Osamu de Sandes Kimura, M.D., Instituto Nacional de Traumatologia e Ortopedia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06554913.0.0000.5273
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Blood Loss, Surgical; Tranexamic Acid Adverse Reaction; Hip Replacement
Keywords: Tranexamic Acid; Blood loss; Tranfusion
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TXA (Experimental): Performed an intravenous bolus administration of 15 mg/kg of TXA to the volunteers after the end of the anesthesia and 15 minutes prior to skin incision.
  Interventions: Drug: Tranexamic Acid Injectable Solution
- Control (Placebo Comparator): This group underwent the same procedures of the TXA group, excepting the preoperative administration of the medication.
  Interventions: Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Solution — Intravenous 15 mg per kilogram tranexamic acid
  Other Names: Lysteda; Transamin
  Arms: TXA
Drug: Placebo - Concentrate
  Arms: Control

SUMMARY:
This study aims to analyze the efficacy of intravenous tranexamic acid (TXA) in patients undergoing total hip arthroplasty (THA).

DETAILED DESCRIPTION:
This was a prospective, experimental, randomized, controlled study of 308 consecutive patients who underwent primary THA from December 2013 to March 2014. 256 volunteers remained in the study, 128 were treated 15 mg/kg intravenous bolus of TXA and 128 did not receive the medication. Participants were followed up at 3 weeks, 3 months, 6 months, 1 year, and then annually after surgery.

The use of TXA resulted in lesser reduction in hemoglobin and hematocrit levels, reduced blood loss, blood transfusion rate, volume of blood products, and stay length even in risk factor patients.

TXA protects risk factor patients against intra and postoperative bleeding and reduces transfusion rates.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who need total hip replacement were included in the initial sample. There was no age limit or restriction regarding gender for admission to the study.

Exclusion Criteria:

* Patients who underwent previous surgery in the same joint, evidence of joint infection, congenital or acquired coagulopathies, active intravascular coagulation, acute occlusive vasculopathy, hypersensitivity to TXA, chronic use of oral and steroid anticoagulants, history of severe or moderate allergy to plasma transfusion, chronic heart disease, malignant neoplasms and autoimmune diseases, patients who needed bone graft or underwent hip arthroplasty revision surgeries, and who did not consent to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin drop | 24 hours post operative
Hematocrit drop | 24 hours post operative
Blood transfusion rate | 5 days
Operative blood loss | 24 hours post operative

SECONDARY OUTCOMES:
Length of stay in hospital | 7 days
Systemic adverse events | 1 year
Thromboembolic efects | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Traumatologia e Ortopedia, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimura OS, Freitas EH, Duarte ME, Cavalcanti AS, Fernandes MB. Tranexamic acid use in high-risk blood transfusion patients undergoing total hip replacement: a randomised controlled trial. Hip Int. 2021 Jul;31(4):456-464. doi: 10.1177/1120700019889947. Epub 2019 Dec 9. PMID 31814452